CLINICAL TRIAL: NCT07246317
Title: A Multicenter, Prospective, Randomized Phase II Trial Evaluating Trastuzumab, Pertuzumab, Docetaxel Combined With QL1706 Versus Combined With Carboplatin as Neoadjuvant Therapy for Early or Locally Advanced HER2+ Breast Cancer
Brief Title: Evaluation of Neoadjuvant Therapy With Trastuzumab, Pertuzumab, Docetaxel, and QL1706 in Early or Locally Advanced HER2+ Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QL-BC-QIBA-1005
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
Keywords: QL1706; HER2+; breast cancer; neoadjuvant therapy; Pertuzumab; Trastuzumab
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Biosimilar Pharmaceuticals; pertuzumab; Docetaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QL1706 arm (Experimental): Trastuzumab, pertuzumab, docetaxel combined with QL1706, q3w, for a total of 4 cycles
  Interventions: Drug: QL1706 injection; Drug: Trastuzumab (or biosimilar); Drug: Pertuzumab (or biosimilar); Drug: Docetaxel
- Standard therapy arm (Active Comparator): Trastuzumab, pertuzumab, docetaxel combined with carboplatin, q3w, for a total of 4 cycles
  Interventions: Drug: Trastuzumab (or biosimilar); Drug: Pertuzumab (or biosimilar); Drug: Docetaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: QL1706 injection — On Day 1 of each cycle at a dose of 5 mg/kg, IV infusion
  Arms: QL1706 arm
Drug: Trastuzumab (or biosimilar) — On Day 1 of each cycle; 8 mg/kg IV loading dose followed by 6 mg/kg IV every 3 weeks
Drug: Pertuzumab (or biosimilar) — On Day 1 of each cycle; 840 mg IV loading dose followed by 420 mg IV every 3 weeks
Drug: Docetaxel — On Day 1 of each cycle at a dose of 75 mg/m², IV infusion
Drug: Carboplatin — On Day 1 of each cycle at a dose of AUC = 4, IV infusion
  Arms: Standard therapy arm

SUMMARY:
This study is a multicenter, prospective, randomized phase II trial designed to observe and evaluate the efficacy and safety of trastuzumab, pertuzumab, docetaxel combined with QL1706 versus combined with carboplatin as neoadjuvant therapy in patients with operable or locally advanced HER2-positive breast cancer.

DETAILED DESCRIPTION:
This multicenter, randomized phase II trial evaluates the efficacy and safety of neoadjuvant therapy with trastuzumab, pertuzumab, and docetaxel plus QL1706 versus the same regimen plus carboplatin in patients with operable or locally advanced HER2-positive breast cancer.

The study will enroll 188 subjects, randomly assigned 1:1 to either the QL1706 combination arm or the carboplatin combination arm, stratified by nodal status and hormone receptor status (<10% vs ≥10%). Both treatment groups will receive four 3-week cycles of assigned therapy followed by surgical resection and response assessment. Postoperative adjuvant treatment will be administered according to investigator discretion and guideline recommendations.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent and compliant.
2. Age 18-70 years.
3. ECOG PS 0-1; life expectancy >6 months.
4. Histologically/cytologically confirmed primary breast cancer.
5. Primary tumor >2cm (by local standard assessment) or node-positive disease.
6. AJCC 8th edition Stage II-IIIC (T2-T4 any N, or any T N1-3 M0) unilateral invasive breast cancer.
7. Confirmed HER2-positive (IHC 3+ or ISH positive). Note: Patients with HER2-negative primary tumor but HER2-positive nodes are eligible.
8. At least one measurable lesion per RECIST 1.1.
9. Agreement to undergo surgery if indicated after neoadjuvant therapy.
10. Willing to provide tumor tissue for biomarker analysis.
11. Adequate organ function:

    * ANC ≥1.5×10⁹/L; PLT ≥100×10⁹/L; HGB ≥90 g/L
    * Albumin ≥30 g/L

      -. TBIL ≤1.5×ULN; ALT/AST ≤2.5×ULN (≤5×ULN if liver metastases); AKP ≤2.5×ULN
    * Creatinine ≤1.5×ULN
    * PT/APTT/INR ≤1.5×ULN (or within therapeutic range if on anticoagulants)
12. For women of childbearing potential: negative pregnancy test within 7 days prior to treatment; must not be breastfeeding.
13. Use of highly effective contraception during and for 3 months after treatment.

Exclusion Criteria:

1. Stage IV metastatic breast cancer or patients deemed ineligible for curative surgery after neoadjuvant therapy.
2. Inflammatory breast cancer.
3. Other malignancies within 3 years, except: those treated with surgery alone and disease-free for 5 years; cured cervical carcinoma in situ, non-melanoma skin cancer, or superficial bladder cancer [Ta, Tis, T1].
4. Prior anti-tumor therapy (chemotherapy, endocrine, anti-HER2) or breast surgery for breast cancer within 3 years (excluding diagnostic biopsy).
5. Major surgery or significant traumatic injury within 28 days before treatment (excluding diagnostic biopsy).
6. Active or history of autoimmune diseases (e.g., autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hypophysitis, vasculitis, nephritis, hyperthyroidism). Exceptions: vitiligo, childhood asthma in complete remission without intervention in adulthood.
7. Current use of immunosuppressants or systemic corticosteroids (>10mg/day prednisone equivalent) within 2 weeks prior to enrollment.
8. History of severe hypersensitivity to monoclonal antibodies.
9. Known central nervous system metastases.
10. Poorly controlled concurrent illnesses, including:

    * Uncontrolled hypertension (SBP>150 or DBP>100 mmHg on medication) or history of hypertensive crisis/encephalopathy.
    * History of heart failure or systolic dysfunction (LVEF <55%).
    * Myocardial ischemia/infarction (≥Grade 2), arrhythmias (QTc≥450ms M, ≥470ms F), or CHF (≥NYHA Class II).
    * Angina requiring medication; clinically significant valvular disease.
    * Active HCV (RNA+), HIV+, syphilis (unless cured), or HBV (HBsAg+ with HBV DNA≥2000 IU/ml or positive qualitative test).
11. Use of Chinese patent medicines with approved anti-tumor indications within 2 weeks prior to treatment.
12. Significant bleeding tendency or clinical bleeding within 3 months; positive fecal occult blood requiring gastroscopy if persistently positive.
13. Tumor invasion or high risk of invasion into major vessels, potentially causing fatal hemorrhage.
14. Pleural, peritoneal, or pericardial effusion requiring drainage (eligible if stable after drainage).
15. Arterial/venous thromboembolic events within 6 months (e.g., CVA, TIA, DVT, PE).
16. Known hereditary or acquired bleeding/thrombotic tendencies (e.g., hemophilia).
17. Severe, non-healing wounds, active ulcers, or untreated fractures.
18. Urinary protein ≥++ confirmed by 24-hour urine protein >1.0g.
19. Active infection, unexplained fever ≥38.5°C within 7 days, or baseline WBC >15×10⁹/L.
20. History of drug abuse or psychiatric disorders.
21. Participation in other anti-tumor drug trials within 4 weeks.
22. Allergy to any study drug or its components.
23. Any condition deemed by the investigator to pose a safety risk or affect study completion.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate using the definition of ypT0/Tis ypN0 (i.e., no invasive residual in breast or nodes; noninvasive breast residuals allowed) at the time of definitive surgery | Up to approximately 16-18weeks
  pCR rate (ypT0/Tis ypN0) is defined as the percentage of participants without residual invasive cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy by current American Joint Committee on Cancer (AJCC) staging criteria assessed by the local pathologist at the time of definitive surgery.

SECONDARY OUTCOMES:
pCR rate using the definition of ypT0/Tis (i.e., no invasive residual in breast or nodes; noninvasive breast residuals allowed) at the time of definitive surgery | Up to approximately 16-18 weeks
  pCR rate (ypT0/Tis) is defined as the percentage of participants without invasive cancer in the breast irrespective of ductal carcinoma in situ or nodal involvement following completion of neoadjuvant systemic therapy by current AJCC staging criteria assessed by the local pathologist at the time of definitive surgery
Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) | Up to approximately 12 weeks
  ORR is defined as the percentage of participants in the analysis population who achieve confirmed complete response (CR: disappearance of all target lesions) or partial response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ.
Event Free Survival | Up to approximately 5 years
  EFS is defined as the time from randomization to any of the following events: preoperative disease progression as determined by the investigator according to RECIST v1.1 - any evidence of contralateral in situ disease is not considered disease progression (PD), while all evidence of contralateral invasive disease is considered PD; postoperative disease recurrence (local, regional, distant, or contralateral); death from any cause. (Whichever occurs first)
Disease-free Survival | Up to approximately 5 years
  DFS is defined as the time from date of surgery (date of no disease) to the first documentation of progressive disease (local, regional, distant, or contralateral) or death.
Overall survival (OS) | Up to approximately 5 years
  OS is defined as the time from randomization to death due to any cause.
Breast-conserving surgery rate | Up to approximately 16-18 weeks
  Breast-conserving surgery rate is the proportion of patients who underwent breast-conserving surgery among all patients who underwent surgery.
Radical resection rate | Up to approximately 16-18 weeks
  The proportion of patients who achieved radical resection among all patients.

OTHER OUTCOMES:
AEs, TRAEs, SAEs | Up to approximately 21-23 weeks
  Incidence and severity of adverse events (AE), treatment-related adverse events (TRAE), serious adverse events (SAE) from cycle 1 day 1 until 30 days post-surgery.

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University (FAH-SYSU), Guangzhou, Guangdong
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Henan University of Science & Technology, Luoyang, Henan
  - Nanyang Central Hospital, Nanyang, Henan
  - The West China Second University Hospital of Sichuan University (WCSUH- SCU), Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Affiliated Hospital of Jiaxing University, Jiaxing, Zhejiang

IPD SHARING:
Plan to Share IPD: No